CLINICAL TRIAL: NCT03472027
Title: A Multicenter Open-Label Single-Arm Multi-Cohort Phase I Study of Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of BCD-145 (JSC BIOCAD, Russia) in Patients With Unresectable/Metastatic Melanoma
Brief Title: Phase I Study of BCD-145 (Anti-CTLA-4) in Patients With Unresectable/Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCD-145-1
Record Dates: First submitted 2018-03-09; First posted 2018-03-21 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BCD-145 Monotherapy Dose Level 1 (Experimental)
  Interventions: Biological: BCD-145
- BCD-145 Monotherapy Dose Level 2 (Experimental)
  Interventions: Biological: BCD-145
- BCD-145 Monotherapy Dose Level 3 (Experimental)
  Interventions: Biological: BCD-145
- BCD-145 Monotherapy Dose Level 4 (Experimental)
  Interventions: Biological: BCD-145
- BCD-145 Monotherapy Dose Level 5 (Experimental)
  Interventions: Biological: BCD-145

INTERVENTIONS:
Biological: BCD-145 — Anti-CTLA-4 monoclonal antibody, IV infusion

SUMMARY:
A Multicenter Open-Label Single-Arm Multi-Cohort Phase I Study of Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of BCD-145 (JSC BIOCAD, Russia) Monotherapy in Patients with Unresectable/Metastatic Melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides a written informed consent and is able to follow the requirements of the Protocol;
2. Age ≥ 18 years
3. Histologically confirmed (well-documented test results; preferably, block specimens available) unresectable (stage III/IV) or metastatic (stage IV) melanoma (the drug will be used as the first of subsequent therapy lines);
4. ECOG score of 0 to 2;
5. Measurable disease (at least one lesion) according to RECIST v1.1 ;
6. Resolved toxicity events from the previous therapy or adverse consequences of surgical interventions to ≤ grade 1 CTCAE v. 4.03, except for chronic/irreversible adverse events not affecting the safety of the study therapy (e.g. alopecia);
7. No severe pathology of organs or systems;
8. Life expectancy of at least 16 weeks from the screening;
9. Patients of childbearing potential enrolled in the study must agree to use reliable contraception methods throughout the study period, beginning 2 weeks before the inclusion in the study and up to 8 weeks after the last dose of BCD-145.

Exclusion Criteria:

1. Severe concomitant illnesses or life-threatening consequences (including pleural/pericardial/peritoneal effusion that requires medical intervention , pulmonary lymphangitis, or involvement of >50% renal parenchyma);
2. Brain metastases ;
3. Severe cardiovascular disorders within 6 months before screening;
4. Autoimmune diseases;
5. Conditions requiring steroids or any other immunosuppressants;
6. Blood disorders: ANC ≤1,500/mm3; platelets ≤100,000/mm3; or Hb ≤90 g/L;
7. Renal function impairment: creatinine ≥1.5 × ULN;
8. Hepatic function impairment: bilirubin ≥1.5 × ULN; AST and ALT ≥2.5 × ULN (5 × ULN for patients with liver metastases), AlkPh ≥ 5 × ULN;
9. Endocrine disorders: abnormal thyroid hormones
10. Prior anticancer treatment within 28 days before starting the study drug (surgery, radiation therapy , or chemotherapy);
11. Known history of more than 6 lines of systemic anticancer chemotherapy (including neoadjuvant and adjuvant CTs);
12. Prior treatment with anti-PD1/PDL1 agents or CTLA4 inhibitors;
13. Concurrent malignancy except for radically resected cervical carcinoma in situ or radically resected basal cell/squamous cell carcinoma;
14. Conditions limiting patient's ability to follow the Protocol requirements (dementia, neurological or psychiatric disorders, drug or alcohol abuse, etc.);
15. Simultaneous participation in any other clinical trial; participation in other clinical trials within 30 days before inclusion in the present study; previous participation in the present study.
16. Acute infections or active chronic infections;
17. Documented hepatitis B, active hepatitis C, HIV or syphilis infection;
18. Intravenous administration of the drug is impossible;
19. Intravenous administration of contrast agents is impossible;
20. Hypersensitivity to any component of BCD-145.
21. Known history of hypersensitivity to monoclonal antibodies;
22. Pregnancy or breastfeeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose-Limiting Toxicities (DLTs) | 85 days
  The Investigators defined Dose-Limiting Toxicities (DLTs) as
  * any treatment-related adverse events of grade 3 or greater,
  * grade 3 or greater immune-mediated toxic effects (defined as an inflammatory process that compromised the function of any organ and was not attributable to another cause) that had the potential to be life threatening with continuation of therapy,
  * immune-mediated toxic effects that did not resolve or improved to grade 2 or less within 14 days of onset

SECONDARY OUTCOMES:
Anti-Drug Antibody levels of BCD-145 | 85 days
  Binding and neutralizing anti-drug antibody levels of BCD-145
Number of Participants With Objective Response | 85 days
  Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
  Pilot efficacy assessment is not the primary objective of this study and will be conducted by surrogate endpoints describing the direct antitumor effect of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Roman A Ivanov, PhD, Study Director — Vice President R&D, JSC BIOCAD
Locations (4):
- Russia (4):
  - N.N. Blokhin National Medical Research Center of Oncology, Moscow
  - JSC "Modern Medical Technologies", Saint Petersburg
  - N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg
  - Saint-Petersburg Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological), Saint Petersburg

IPD SHARING:
Plan to Share IPD: No